CLINICAL TRIAL: NCT02697448
Title: Comparison of Propofol and Sevoflurane as a Primary Anesthetic for Cardiac Ablation of Atrial Fibrillation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, George Guldan, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00044072
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator): Participants receiving propofol as anesthetic for cardiac ablation.
  Interventions: Drug: propofol
- sevoflurane (Active Comparator): Participants receiving sevoflurane as anesthetic for cardiac ablation.
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — Participant receives propofol as anesthetic for cardiac ablation.
  Arms: propofol
Drug: sevoflurane — Participant receives sevoflurane as anesthetic for cardiac ablations.
  Arms: sevoflurane

SUMMARY:
Comparison of propofol and sevoflurane as a primary anesthetic for cardiac ablation of atrial fibrillation

DETAILED DESCRIPTION:
A side effect of some volatile anesthetics, such as isoflurane and desflurane, is enhanced automaticity, accounting for secondary atrial pacemakers. Volatile anesthetics also have varying effects on the AV node and His-Pukinje system. These agents also prolong the QT interval and, for this reason, volatile anesthetics as a group have at times been avoided for atrial fibrillation ablation due to the fear that they may affect the efficacy of the ablation and increase recurrence. However, sevoflurane does not have the effects shown for other volatile anesthetics cardiac conduction. At this point there has not been a study comparing propofol, a non volatile anesthetic typically used in these cases, to sevoflurane, a volatile anesthetic, to determine if volatile anesthetics should be avoided during these procedures. This study will challenge the existing belief that sevoflurane increases the length of time to ablate atrial fibrillation and also decreases the efficacy of the ablation.

ELIGIBILITY:
Inclusion Criteria:

* have paroxysmal atrial fibrillation
* undergoing their first ablation.

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George J Guldan, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Sevoflurane
Started | 67 | 68
Completed | 62 | 63
Not Completed | 5 | 5
Not completed — Protocol Violation | 2 | 4
Not completed — Clinical concerns during ablation | 1 | 1
Not completed — No data collected | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Sevoflurane | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.63) | 64.3 (11.3) | 66.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 46 | 49 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 58 | 113
  Black, or Other | 7 | 5 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (5.81) | 30.8 (7.08) | 30.6 (6.42)

OUTCOME MEASURES:

1. Primary Outcome: Procedure Duration
Description: The duration of the procedure in minutes.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
minutes | 159.2 [145.5 to 172.9] | 170.7 [158.1 to 183.3]

2. Primary Outcome: Time to Extubation
Description: The time from procedure end to the time the patient is extubated, in minutes. A longer extubation time is a worse outcome.
Time Frame: Procedure end time to time of extubation
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
Minutes | 11 [6.0 to 15] | 8 [4.0 to 12.0]

3. Other Pre Specified Outcome: Post-Operative Pain
Description: Post-Operative Pain was measured on a Numeric Rating Scale of 0-10, and assessed on Post-Op Day 1 by asking the patient to rate their pain while resting. Zero meant no pain, and 10 meant worst pain imaginable. A higher number is a worse outcome.
Time Frame: Post-Op Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
units on a scale | 2 [1 to 4] | 2 [1 to 4]

4. Other Pre Specified Outcome: Number of Participants With Post-Operative Nausea and Vomiting
Description: On Post-Op Day 1, patients were asked if they had experienced any nausea of vomiting since their procedure by answering "yes" or "no".
Time Frame: Time of procedure end to post-op day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
Participants | 4 | 4

5. Other Pre Specified Outcome: Post-Operative Alertness
Description: Patients were asked on Post-Op Day 1 to rate how alert they felt on a numeric rating scale from 0-10. Zero meant very groggy, and 10 meant back to normal alertness. The higher the number, the better the outcome.
Time Frame: Post-Op Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
units on a scale | 9 [7 to 10] | 9 [7 to 10]

6. Other Pre Specified Outcome: Incidence of Atrial Fibrillation
Description: This outcome examines the association between treatment group and postoperative time with recurrence of atrial fibrillation in the first 6 months following the procedure. The numbers reported reflect whether or not the participant experienced an atrial fibrillation in the specified time period.
Time Frame: 2 weeks post-op, 3 months post-op, and 6 months post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Sevoflurane
Number analyzed (Participants) | 62 | 63
Participants
  2 weeks post-op | 13 | 12
  3 months post-op | 12 | 18
  6 months post-op | 10 | 17

ADVERSE EVENTS:
Time Frame: Adverse events related to the study intervention were collected from the time randomization occurred and the intervention was administered, and 24 hours post-operatively.
Arm/Group | Propofol | Sevoflurane
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 4/62 | 4/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=62) | Sevoflurane (N=63)
Post-Operative Nausea and/or Vomiting (Nervous system disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT02697448/Prot_SAP_000.pdf